CLINICAL TRIAL: NCT03317262
Title: Multi-center, Open, Non-invasive, Prospective, Clinical Observational Study in Patients in Greece With Depression and Generalized Anxiety Disorder Treated With Sitalopram and Not Satisfactorily Controlled.
Brief Title: Prospective Study of the Evaluation of Disease contRol and the Quality of Life of Patients With depressiOn and With or Without aNxiety disOrders in the Greek populatIon
Acronym: PRONOI
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-CTL-EL-76
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2018-03

CONDITIONS: Depression; Anxiety Disorders
Keywords: quality of life, citalopram, quetiapine, pregabalin
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Depression is a psychiatric disorder that affects mood, thoughts and is usually accompanied by physical annoyances. It affects the person's eating habits, his sleep, the way he sees himself and the way he thinks and understands. Depressed emotion has great tension, lasts longer and leads to a reduction in the person's functioning in many areas of his life.

Generalized Anxiety Disorder (GAD) is the psychiatric disorder characterized by a multitude of diverse organic responses as well as a generalized, persistent and indeterminate anxiety that covers almost all of the individual's activities. It is a diffuse and intense negative mood and anxiety that is present for most of the day and whose exact causes are often undetectable.

DETAILED DESCRIPTION:
The Hamilton Depression Scale is the most widely used scale for measuring the severity of depression worldwide. It was designed to measure the severity of depression in already diagnosed patients with major depressive disorder. It includes 17 entries rated from 0 to 2 or from 0 to 4, thus giving a total score ranging from 0-50.

The scores are scored through the symptoms reported by the patient during the interview, the evaluator's observations and the information collected from third parties (relatives, nurses). The markings do not distinguish between the intensity and frequency of the symptoms, but these two should be equally at the discretion of the assessor. The scale covers the condition of the patient in the week preceding the mark for most symptoms, except for sleep disorders related to the last three days.Health-related quality of life is calculated using weighted questionnaires focusing on the general health level of the individual or the impact of specific diseases on the quality of life of the patient.

These questionnaires are based on a common theoretical background, according to which the measurement of biological functionality is a basic, but not sufficient, assessment of health. Apart from the good functioning of organic systems, which represents the traditional biomedical model of health, the need for an assessment of the general well-being and functioning of the individual in all areas of his life is also important.

The EQ-5D questionnaire is a self-completed tool for measuring the quality of life and consists of two parts:

The first part records the person's health profile. Five dimensions are used, referring to (a) mobility, (b) self-handling, (c) routine activities, (d) pain-discomfort and (e) stress-depression. Each of these dimensions takes three values: 1 = no problem, 2 = some problems, 3 = significant problems. Altogether, three health situations are recorded, representing 243 cases. The best mental state is described as "11111", meaning that there is no problem in terms of mobility, self-care, routine activities, pain and anxiety. The worst mental health status gets the "33333" values, which means significant problems in the above five dimensions.

The second part presents a visual analogue scale (VAS) in the form of a "health thermometer", which takes values from 0 = worse mental health to 100 = excellent mental health. Intermediate values of the optical proportional scale indicate intermediate health status. This scale is based on the person's subjective assessments of his / her state of health.

Using the EQ-5D, it is possible to estimate the benefit enjoyed by the individual from different health situations.

The HAM-A scale was one of the first assessment scales developed to measure the severity of anxiety symptoms and is still used up to now in both clinical and research environments.

The scale consists of 14 elements, which are determined by a series of symptoms, and measures both mental (mental stimulation and psychological discomfort as well as physical anxiety (physical anxiety disorders).

Each question is scored on a scale of 0 (none) to 4 (very serious), with a total score of 0 to 56. A score of less than 17 indicates mild severity, 18-24 mild to moderate severity and 25-30 mild to severe.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Male or female asthma patients over 18 years of age
* Compliance with treatment
* Compliance with study procedures
* Patients already receiving or to receive citalopram
* Patients not adequately controlled by citalopram
* Patients not adequately controlled by citalopram and at the same time having a generalized anxiety disorder
* Patients not regulated at all

Exclusion Criteria:

* Unsigned patient consent
* Male or female asthma patients under 18 years of age
* Non-compliance with treatment
* Non-compliance in study procedures
* Patients who do not meet the Product SmPC criteria
* Patients receiving MAO inhibitors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with depression and anxiety disorders
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Disease Control | 6 months
  Change in HAM-D scale
  The Hamilton Depression Scale is the most widely used scale for measuring the severity of depression worldwide. It was designed to measure the severity of depression in already diagnosed patients with major depressive disorder. It includes 17 entries rated from 0 to 2 or from 0 to 4, thus giving a total score ranging from 0-50.
Disease Control | 6 months
  Change in HAM-A scale The HAM-A scale was one of the first assessment scales developed to measure the severity of anxiety symptoms and is still used up to now in both clinical and research environments.
  The scale consists of 14 elements, which are determined by a series of symptoms, and measures both mental (mental stimulation and psychological discomfort as well as physical anxiety (physical anxiety disorders).
  Each question is scored on a scale of 0 (none) to 4 (very serious), with a total score of 0 to 56. A score of less than 17 indicates mild severity, 18-24 mild to moderate severity and 25-30 mild to severe.

SECONDARY OUTCOMES:
Quality of Life | 6 months
  Change in EuroQol-5D scale
  The EQ-5D questionnaire is a self-completed tool for measuring the quality of life and consists of two parts:
  The first part records the person's health profile. Five dimensions are used, referring to (a) mobility, (b) self-handling, (c) routine activities, (d) pain-discomfort and (e) stress-depression. Each of these dimensions takes three values: 1 = no problem, 2 = some problems, 3 = significant problems. Altogether, three health situations are recorded, representing 243 cases. The best mental state is described as "11111", meaning that there is no problem in terms of mobility, self-care, routine activities, pain and anxiety. The worst mental health status gets the "33333" values, which means significant problems in the above five dimensions.

CONTACTS AND LOCATIONS:
Locations (1):
- Private Office, Larissa, Greece